CLINICAL TRIAL: NCT01427088
Title: Short-Term Response of Serum Brain-Derived Neurotrophic Factor to Repetitive Transcranial Magnetic Stimulation in Patients With Chronic Schizophrenia
Brief Title: rTMS-induced Cumulative Pattern of sBDNF in Chronic Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeonbuk Provincial Maeumsarang Hospital (Other)
Responsible Party: Principal Investigator, HWANG TAEYOUNG, Director, Insan Research Center for Psychiatry, Jeonbuk Provincial Maeumsarang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: rTMS-sBDNF-SPR-2011
Record Dates: First submitted 2011-08-28; First posted 2011-09-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: rTMS-induced cumulative pattern of sBDNF
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- repetitive TMS (Experimental): repetitive TMS is a quantified stimulation method of specifie area of brain, for which CR Technology, TAMAS for repetitive TMS was used.
  Interventions: Device: CR Technology, TAMAS for repetitive TMS

INTERVENTIONS:
Device: CR Technology, TAMAS for repetitive TMS — repetitive TMS, lef DLPFC, 20Hz, 100% of MEP, 2weeks

SUMMARY:
This study aims at investigating the neuroplastic potential and the possible factors affecting rehabilitation in chronic schizophrenia patients on stable medication, by investigating the cumulative pattern of serum BDNF representing the neuroplasticity in the brain, through quantitative stimulus such as rTMS.

DETAILED DESCRIPTION:
Subjects who have been enrolled for this study will take baseline evaluation for sociodemographic data and serum level of BDNF, plasma Prolaction, and magnesium, etc. And then, weekday regular stimulation through rTMS will be applied on DLPFC of brain. After the completion of stimulation for 2 weeks, the change or response of serum BDNF will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* duration of illness over 10 years
* on stable medication, antipsychotics
* no change on medication within at least 2 weeks
* Diagnosis of Schizophrenia according to DSM-IV-TR

Exclusion Criteria:

* left or both-handedness
* anticonvulsant use
* lorazepam equivalent over 3 mg

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
change from baseline of serum BDNF concentration | baseline-1 week-2 week-4 week

CONTACTS AND LOCATIONS:
Overall Officials: TAEYOUNG HWANG, M.D., M.P.H., Principal Investigator — Jeonbuk Provincial Maeumsarang Hospital
Locations (1):
- Jeonbuk Provincial Maeumsarang Hospital, Wanju, Jeollabuk-do, South Korea